CLINICAL TRIAL: NCT04925700
Title: The Oral Microbiome in Oral Squamous Cell Carcinoma
Brief Title: The Oral Microbiome in OSCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, David R. Drake, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202012278
Record Dates: First submitted 2021-05-27; First posted 2021-06-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Lozenge (Experimental)
  Interventions: Dietary Supplement: ProDentis Lozenge
- Placebo Lozenge (Placebo Comparator)
  Interventions: Other: Placebo Lozenge

INTERVENTIONS:
Dietary Supplement: ProDentis Lozenge — 1-2 ProDentis Lozenges per day
  Arms: Probiotic Lozenge
Other: Placebo Lozenge — 1-2 Placebo Lozenges per day
  Arms: Placebo Lozenge

SUMMARY:
Previous work by a number of scientific teams has revealed that the types of bacteria that colonize the mouth differ between health and pre-cancerous or cancerous oral lesions. The purpose of this study is to investigate the extent of these changes and to correlate the changes with alterations in the activities of the host's own oral tissues. In doing so, we believe we can gain a better understanding of how particular bacterial species, or consortia of species, can result in an individual having an increased risk of the most common type of oral cancer -- oral squamous cell carcinoma. This knowledge may also lead to the identification of salivary biomarkers that can be used for clinical evaluation or screening. In addition, we seek to determine the extent to which a probiotic regimen can help prevent or rectify the disease-related changes in the types of bacterial colonizing the mouth. The microbiome in health, pre-cancerous lesions, and cancerous lesions will be determined from remnant microbial DNA in banked tissue samples. The effects of probiotics on the oral microbiome will be determined from DNA collected from swabs of oral tissue at baseline and then after 3 to 6 months of probiotic usage.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (21-70 years old) who have been diagnosed with oral dysplasia or that have been treatment-planned as wait and watch or
2. Adults (21-70 years old) or who have been diagnosed with oral squamous cell carcinoma, or matched healthy controls free of any oral lesions

Exclusion Criteria:

1. Adults who have had a course of antibiotics that was completed less than 3 months prior to the study;
2. Adults with any immunosuppressive condition or medication that would put the subject at risk of consuming daily probiotics;
3. Adults who regularly use probiotic dietary supplements
4. Adults that have alcohol/tobacco use history that does not match study population - this if for the healthy controls arm only.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in the oral microbiome composition over time | Up to 3 months
  16S Genomic Profiling will be done in all recruited subjects via oral swab of pre-cancerous or cancerous oral lesion
Determine the Effect of ProDentis on the Oral Microbiome | Up to 3 months
  Pre-Cancerous lesion is treatment planned as "watch-and-wait" or oral lesion is not present, recruited subjects will be randomly assigned to either the probiotic lozenge or placebo lozenge group.

CONTACTS AND LOCATIONS:
Overall Officials: David Drake, MS, PhD, Principal Investigator — University of Iowa College of Dentistry
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States